CLINICAL TRIAL: NCT06296498
Title: The Effect of Application of L-PRF in Periodontal Surgery on Clinical Parameters and Patient Related Outcome Measures: A Randomized, Controlled, Clinical Study.
Brief Title: Application of L-PRF in Periodontal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20230505HU
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Periodontal Diseases
Keywords: Open flap debridement; Periodontal surgery; Periodontal wound healing
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: The proposed study is a split-mouth design, randomized, prospective clinical trial in which we will use either OFD alone or OFD + L-PRF for periodontal surgery. Both procedures are standard of care
Who Masked: Participant
Masking Description: Participants will be blinded to the intervention which they are randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group OFD + L-PRF (Active Comparator): Open flap debridement (OFD) with L-PRF is used during periodontal surgical procedure that is used to improve periodontal health by providing access to the tooth roots and alveolar bone.
  Interventions: Procedure: Leukocyte Platelet-rich fibrin
- Group OFD (Other): Open flap debridement (OFD) is one periodontal surgical procedure that is used to improve periodontal health by providing access to the tooth roots and alveolar bone.
  Interventions: Other: Standard of care OFD

INTERVENTIONS:
Procedure: Leukocyte Platelet-rich fibrin — Leukocyte-PRF (L-PRF) contains neutrophils and macrophages that facilitate bacteria and necrotic tissue elimination via phagocytosis
  Other Names: L-PRF
  Arms: Group OFD + L-PRF
Other: Standard of care OFD — Open flap debridement (OFD) is one periodontal surgical procedure that is used to improve periodontal health by providing access to the tooth roots and alveolar bone.
  Other Names: Open Flap Debridement
  Arms: Group OFD

SUMMARY:
The study will compare the clinical outcomes of the two procedures, open flap debridement (OFD) compared to open flap debridement with leukocyte and platelet-rich fibrin (L-PFR) as well as differences in patient postoperative pain perception.

DETAILED DESCRIPTION:
Randomization to one of two standard of care procedures:

1. Test group: After gingival flap reflection and debridement of bone and root surfaces L-PRF will be applied to the alveolar bone, tooth roots, and gingival flap prior to suturing.
2. Control group (Standard of care): Gingival flap reflection and debridement of bone and root surfaces, followed by suturing of the gingival flaps.

The study is a split-mouth design, randomized, prospective clinical trial. The protocol will randomize gingival quadrants in subjects to one of two standard of care procedures OFD or OFD + L-PRF. Patients needing periodontal surgery to correct periodontal disease will be enrolled. There will be two subject groups in this study. Each subject will be randomized to one of the treatments for the first quadrant and the contralateral quadrant will receive the other treatment. No risk is expected from being assigned to either group as both procedures are standard of care, with possible benefit of enhanced wound healing and bone regeneration in the test group.

Allocation of subjects into test group or control group will be based on numbers drawn from a stack of sealed envelopes.

ELIGIBILITY:
Inclusion Criteria:

* Patients between age 18 and 89
* Patients needing open flap debridement procedures for periodontal disease in one or more teeth in the same arch bilaterally (split mouth)
* Patients must be nonsmokers, former smokers, or current smokers who smoke <10 cigarettes per day, by self-report
* Female patients to include non- pregnant women of child-bearing potential.

Exclusion Criteria:

* Patients who disclose that they will not be able to cooperate with the follow-up schedule.
* Patients who are mentally incompetent, prisoners, or pregnant (as obtained via chart review or self-report)
* Pregnant women or women intending to become pregnant during the study period
* Smokers who smoke > 10 cigarettes per day

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-08-19 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
Probing depth | 3 months and 6 months
  Depth of gingival pocket
Postoperative Pain (PROM) | 12 to 168 hours post surgery
  Change in Patient reported outcome measures measured by a 10 point scale with 0 being no pain and 10 is the worst pain ever experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Powell, DDS, MS, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All deidentified participant data will be shared with colleagues
Supporting Information: Study Protocol, SAP
Time Frame: After study completion in a peer review journal